CLINICAL TRIAL: NCT03705546
Title: The Impact of Physical Activity on the Postoperative Symptoms, Complications, and Quality of Life Among Lung Cancer Survivors: A Prospective Cohort Study
Brief Title: The Impact of Physical Activity on the Postoperative Symptoms, Complications, and Quality of Life Among Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC 2015-11-025-002(C)
Record Dates: First submitted 2018-10-05; First posted 2018-10-15 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine the impact of physical activity on the postoperative symptoms, complication, and quality of life.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) survivor is increasing as developing early diagnosis and perioperative management. Despite multidisciplinary treatment, Surgery is the primary treatment option for cure in NSCLC. The patients with lung cancer who underwent surgery have limitation of pulmonary function and high risk of co-morbidities. Perioperative physical activity has been shown to reduce symptoms and prevent complications, improve long term quality of life after surgery. But validated exercise regimen has not been established for lung cancer patients. Therefore, Evidence-based guideline focusing on lung cancer after surgery is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with lung cancer
* Patients who are able to walk with ECOG (Eastern Cooperative Oncology Group) performance status < 1
* Patients who understand the purpose of this study and provide the written informed consent

Exclusion Criteria:

* Patients who have difficulty for walking
* Patients with history of other cancer in the last 3 years
* Patients with neoadjuvant chemotherapy and/or radiation therapy
* Patients who are diagnosed with recurrent lung cancer or multiple cancer
* Foreigner of patients from overseas who are not able regularly participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population in this study consists of patients who are diagnosed with lung cancer and scheduled for surgery in a lung cancer center at Seoul.
Sampling Method: Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
The change of quality of life: (EORTC QLQ) core30 (C30) | Before surgery (baseline), and 1, 6, 12, 24, 36, 48, and 60 months after surgery
  The change of quality of life is measured using the European Organization for Research Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) core30 (C30). The scale for quality of life is transformed into a score from 0 to 100, derived by 4-point Likert scale. A higher score represents a higher level of quality of life.

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Within 30 days after surgery
  Incidence of pulmonary complications including air leak, atelectasis, pleural effusion, pneumonia, etc.
The change of symptom | Before surgery (baseline), and 1, 6, 12, 24, 36, 48, and 60 months after surgery
  The change of symptom is measured using the European Organization for Research Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) lung cancer module 13 (LC13). The scale for symptom is transformed into a score from 0 to 100, derived by 4-point Likert scale. A higher score represents a higher level of symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kwan Kim, Ph.D., Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong S, Shin S, Jeon YJ, Lee G, Cho JH, Kim HK, Shim YM, Cho J, Kang D, Park HY. Factors associated with failure of cardiopulmonary function recovery after lung cancer surgery. Respirology. 2023 Nov;28(11):1060-1068. doi: 10.1111/resp.14581. Epub 2023 Aug 29. PMID 37642118
- [Derived] Shin S, Kong S, Kang D, Lee G, Cho JH, Shim YM, Cho J, Kim HK, Park HY. Longitudinal changes in pulmonary function and patient-reported outcomes after lung cancer surgery. Respir Res. 2022 Aug 30;23(1):224. doi: 10.1186/s12931-022-02149-9. PMID 36042472
- [Derived] Lee H, Kim HK, Kang D, Kong S, Lee JK, Lee G, Shin S, Cho J, Zo JI, Shim YM, Park HY. Prognostic Value of 6-Min Walk Test to Predict Postoperative Cardiopulmonary Complications in Patients With Non-small Cell Lung Cancer. Chest. 2020 Jun;157(6):1665-1673. doi: 10.1016/j.chest.2019.12.039. Epub 2020 Jan 25. PMID 31987880